CLINICAL TRIAL: NCT00804336
Title: Phase I Study of Pasireotide (SOM230) in Combination With RAD001 in Patients With Advanced Neuroendocrine Tumors
Brief Title: Pasireotide in Combination With RAD001 in Patients With Advanced Neuroendocrine Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Jennifer Chan, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-087
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Neuroendocrine Tumor; Carcinoid Tumor; Pancreatic Neuroendocrine Tumor
Keywords: pasireotide; SOM230; RAD001
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Adenoma, Islet Cell | interventions — pasireotide; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pasireotide and RAD001 (Experimental): RAD001 was administered orally as a once-daily dose. Pasireotide s.c. was self-administered s.c. twice daily for 4 weeks. If pasireotide s.c. was tolerated, patients received pasireotide LAR i.m. at the corresponding dose level. Pasireotide s.c. was continued for an additional 2 weeks after administration of pasireotide LAR until anticipated steady-state levels of pasireotide LAR were achieved. Pasireotide LAR was administered every 28 days. Cycles for everolimus and pasireotide LAR were repeated every 28 days.
  Interventions: Drug: SOM230; Drug: RAD001

INTERVENTIONS:
Drug: SOM230 — Given subcutaneously twice a day for four weeks then given intramuscularly once every four weeks thereafter
  Other Names: pasireotide
Drug: RAD001 — Given orally once a day

SUMMARY:
The purpose of this research study is to determine the safety of the combination of SOM230 and RAD001, as well as determine the highest dose of this combination that can be given to people safely. SOM230 is an investigational drug that is similar to Sandostatin LAR. Sandostatin is an approved drug for the use of treating symptoms of neuroendocrine tumors. SOM230 has shown to be effective in patients who have become resistant to Sandostatin and may also stop cancer cells from growing. RAD001 is an investigational drug that also may stop cancer cells from growing.

DETAILED DESCRIPTION:
* Participants will be receiving two study medications, SOM230 and RAD001, during each treatment cycle. Each treatment cycle lasts 4 weeks.
* For the first four weeks of treatment, the participant will self-administer the SOM230 twice a day by subcutaneous injection. If they tolerate the SOM230 after 4 weeks, they will switched to the long-acting SOM230 which will be administered during scheduled treatment visits once every 4 weeks. For the first two weeks after switching to the long-acting SOM230, participants will continue to self-administer the short-acting SOM230 twice a day.
* RAD001 will be taken orally once every day.
* On Day 1 of every cycle, a physical exam and blood tests will be performed. Following every 2 cycles of treatment an assessment of the tumor by CT scan wil be performed.
* Pharmacokinetic (pK) blood samples will be taken on days 1 and 15 of cycle one. The pK samples will be taken right before the study drug is administered and then 1, 2, 3, and 5 hours later.

ELIGIBILITY:
Inclusion Criteria:

* Locally unresectable or metastatic neuroendocrine tumor. Patients must have confirmed low-grade or intermediate-grade neuroendocrine carcinoma. Patients with poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoid, and small cell carcinoma are not eligible.
* 18 years of age or older
* Minimum of four weeks since any major surgery, completion of radiation, of completion of all prior systemic anticancer therapy.
* ECOG Performance Status 0,1, or 2.
* Life expectancy 12 weeks or more.
* Adequate bone marrow, liver and renal function as outlined in the protocol
* Negative serum pregnancy test for women of childbearing potential.
* Fasting serum cholesterol less than or equal to 300mg/dL or less than or equal to 7.75mml/L AND fasting triglycerides of less than or equal to 2.5 x ULN.

Exclusion Criteria:

* Chronic treatment with systemic steroids or another immunosuppressive agent.
* Immunization with attenuated live vaccines during study or within 1 week of study entry.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Prior or concurrent malignancy, except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years.
* Uncontrolled diabetes mellitus or a fasting plasma glucose of > 1.5 ULN.
* Symptomatic cholelithiasis
* Congestive heart failure, unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment.
* Presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result.
* Any severe and/or uncontrolled medical condition or other conditions that could affect their participation in the study such as: severely impaired lung function; active or uncontrolled infection/disorders; nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by treatment with the study therapy; impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001; history of alcohol or drug abuse in the 6 month period prior to receiving treatment.
* Known hypersensitivity to RAD001 or other rapamycins or its excipients.
* Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR or s.c. formulations.
* History of non-compliance to medical regimens.
* Patients taking medication known to inhibit, induce, or be a substrate to isoenzyme CYP3A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2014-09 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose for pasireotide (SOM230) in combination with RAD001 in this patient population. | 2 years
To determine the dose-limiting toxicities of the combination in this patient population. | 2 years

SECONDARY OUTCOMES:
To determine the pharmacokinetics of combined treatment | 2 years
To make a preliminary assessment of the anti-tumor activity of the combination in this patient population | 2 years
To determine the objective response rate | 3 years
To determine the duration of response | 3 years
To determine the progression free survival and overall survival of patients receiving this combination. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ang Chan, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Chan JA, Ryan DP, Zhu AX, Abrams TA, Wolpin BM, Malinowski P, Regan EM, Fuchs CS, Kulke MH. Phase I study of pasireotide (SOM 230) and everolimus (RAD001) in advanced neuroendocrine tumors. Endocr Relat Cancer. 2012 Sep 14;19(5):615-23. doi: 10.1530/ERC-11-0382. Print 2012 Oct. PMID 22736724